CLINICAL TRIAL: NCT00794690
Title: Influence of Black Cohosh (Cimicifuga Racemosa) Use by Postmenopausal Women on Total Hepatic Perfusion and Liver Functions
Brief Title: Safety Study of Black Cohosh Use by Postmenopausal Women on the Liver
Acronym: CR-LIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Prof. Ezat Hamed Sayed, Department of Obstetrics & Gynecology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR and the liver
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Menopause
Keywords: cimicifuga racemosa; liver blood flow and functions
MeSH Terms: interventions — black cohosh root extract; Klimadynon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- black cohosh extract, liver (Experimental): 100 postmenopausal women
  Interventions: Drug: Cimicifuga racemosa extract for the group

INTERVENTIONS:
Drug: Cimicifuga racemosa extract for the group — 40 mg of Cimicifuga racemosa extract daily dor 12 months
  Other Names: Klimadynon®

SUMMARY:
Black Cohosh extract is a form of phytoestrogen (estrogen of plant origin) that is effective in controlling bothersome hot flushes, while avoiding the dangers of using hormones. Recent case reports pointed to potential toxicity of black cohosh on the liver. The investigators are trying to verify or refute such allegations.

DETAILED DESCRIPTION:
The aim of this prospective longitudinal clinical trial is to evaluate changes in total hepatic blood flow and liver functions among postmenopausal women using black cohosh (cimicifuga racemosa) extract for twelve consecutive months for relief of vasomotor symptoms.

Prior to using a daily dose of 40 mg of a dry extract preparation of cimicifuga racemosa (Klimadynon®) and twelve months after, total hepatic blood flow will be assessed by color Doppler ultrasound. Moreover, prothrombin time & concentration, serum albumin, bilirubin, gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* an age over 40 years
* with a lapse of one year after the last menstruation
* symptomatic women without gynecological illness
* after naturally occurring menopause
* had never used hormonal therapy or had stopped using them for >6 months
* accepting to participate after receiving adequate description of the study
* accessible for regular follow-up.

Exclusion Criteria:

* vaginal bleeding
* active or chronic liver disease and /or abnormal liver functions
* present or past thromboembolic disease
* present or past neoplasia of the breast or uterus
* an endometrial thickness >5 mm by TVS
* use of alternative or complementary medicines or herbs for menopausal symptoms within the previous three months

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Effect on hepatic perfusion and liver functions | 12 months

SECONDARY OUTCOMES:
Efficacy and tolerability | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: AHMED M NASR, MD, Principal Investigator — ASSIUT UNIVERSITY, EGYPT
Locations (1):
- Dept. Obstetrics and Gynecology, Assiut University, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Mahady GB, Low Dog T, Barrett ML, Chavez ML, Gardiner P, Ko R, Marles RJ, Pellicore LS, Giancaspro GI, Sarma DN. United States Pharmacopeia review of the black cohosh case reports of hepatotoxicity. Menopause. 2008 Jul-Aug;15(4 Pt 1):628-38. doi: 10.1097/gme.0b013e31816054bf. PMID 18340277
- [Background] Chow EC, Teo M, Ring JA, Chen JW. Liver failure associated with the use of black cohosh for menopausal symptoms. Med J Aust. 2008 Apr 7;188(7):420-2. doi: 10.5694/j.1326-5377.2008.tb01691.x. No abstract available. PMID 18393750